CLINICAL TRIAL: NCT07000968
Title: The Effect of Task-Oriented Training and Virtual Reality Training on Balance, Gait and Fatigue in Individuals With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1421
Record Dates: First submitted 2024-02-08; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis; Balance Impairment, Gait Disorders, Fatigue; Multiple Sclerosis Bening; Multiple Sclerosis Relapsing Remitting
Keywords: Task Oriented Training; Virtual Reality; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Mobility Limitation; Fatigue; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group, interventional study including two active intervention arms. Participants remain in their assigned group for the duration of the study.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Virtual Reality Training Group (Experimental): Virtual Reality Training Procedure; In general, virtual reality training will be developed taking into account neurorehabilitation principles; Type of game and specificity (there will be exercises specific to the disease), Intensity (will be gradually increased), Progress (exercises will be gradually progressed, variability (the environment will be changed) and Feedback (visual and auditory feedback will be provided). The virtual reality training to be applied will also be fun, It will include attention and problem-solving ability. The difficulty and skill level will gradually increase in order to ensure continuity of motivation and motor learning in individuals. It will be aimed to perform the exercises at moderate to severe intensity. The intensity level of the exercises will be at moderate intensity, and the perceived effort according to the Borg Scale will be 12- It will be checked by asking for 15 points.
  Interventions: Other: Virtual Reality Training Group
- Conventional Training Group (Other): Individuals in this group will continue classical physiotherapy exercises. There will be no intervention by us in the traditional training group.
  Interventions: Other: Conventional Training Group
- Task-Oriented Training Group (Experimental): Task Oriented Training Procedure; Task-oriented training focusing on improving balance and walking will consist of 8 different exercise stations. Individuals will continue the exercise at each station for 4 minutes and rest for 1 minute before moving on to the next station. The training completed in this way will consist of a total of 40 minutes and the exercise stations will be applied following the determined order: The exercises will first be demonstrated by the physiotherapist. The aim is to perform exercises at moderate to vigorous intensity. It will be checked that the intensity level of the exercises is moderate and that the perceived effort is 12-15 points according to the Borg Scale. Perception of perceived exertion; It will be controlled by asking to increase the speed, changing the ground, giving double tasks and using obstacles made of wooden blocks. Individuals will be given visual and auditory positive feedback during the exercises.
  Interventions: Other: Task-Oriented Training Group

INTERVENTIONS:
Other: Virtual Reality Training Group — Virtual Reality Training Procedure; In general, virtual reality training will be developed taking into account neurorehabilitation principles; Type of game and specificity (there will be exercises specific to the disease), Intensity (will be gradually increased), Progress (exercises will be gradually progressed, variability (the environment will be changed) and Feedback (visual and auditory feedback will be provided). The virtual reality training to be applied will also be fun, It will include attention and problem-solving ability. The difficulty and skill level will gradually increase in order to ensure continuity of motivation and motor learning in individuals. It will be aimed to perform the exercises at moderate to severe intensity. The intensity level of the exercises will be at moderate intensity, and the perceived effort according to the Borg Scale will be 12- It will be checked by asking for 15 points.
  Arms: Virtual Reality Training Group
Other: Task-Oriented Training Group — ask Oriented Training Procedure; Task-oriented training focusing on improving balance and walking will consist of 8 different exercise stations. Individuals will continue the exercise at each station for 4 minutes and rest for 1 minute before moving on to the next station. The training completed in this way will consist of a total of 40 minutes and the exercise stations will be applied following the determined order: The exercises will first be demonstrated by the physiotherapist. The aim is to perform exercises at moderate to vigorous intensity. It will be checked that the intensity level of the exercises is moderate and that the perceived effort is 12-15 points according to the Borg Scale. Perception of perceived exertion; It will be controlled by asking to increase the speed, changing the ground, giving double tasks and using obstacles made of wooden blocks. Individuals will be given visual and auditory positive feedback during the exercises.
  Arms: Task-Oriented Training Group
Other: Conventional Training Group — Individuals in this group will continue classical physiotherapy exercises. There will be no intervention by us in the traditional training group.
  Arms: Conventional Training Group

SUMMARY:
Introduction: Multiple sclerosis (MS) is a chronic disease of the central nervous system. Task-focused training is an approach that relies on multiple repetitions of motor performance. Virtual reality is a technology that combines computer graphics to create a realistic world that responds to the user's responses.

Purpose: The study was planned to observe the effect of virtual reality training on balance, walking and fatigue and to compare it with task-oriented training.

Materials and Methods: The study, designed as a randomized controlled study, will include individuals with multiple sclerosis between the ages of 20-65. The population of the study consists of individuals with MS at Elazig Private Ada Special Education and Rehabilitation Center. Individuals who agree to participate in the study and meet the inclusion criteria will be selected by trying to reach the entire relevant population and will be divided into three groups using the sealed envelope method. Individuals will be evaluated before treatment and at the 8th week after treatment. One of the experimental groups will receive task-oriented training in the clinic 3 days a week, 40 minutes a day for 8 weeks, virtual reality training will be applied to the other, and conventional training will be applied to the control group. Expanded disability status scale to evaluate physical disability; balance assessment berg balance scale; gait assessment rivermead visual gait assessment scale; Fatigue assessment will be evaluated using the fatigue severity scale.

Result: The effects of task-oriented and virtual reality training groups on balance, walking and fatigue will be interpreted by comparing the evaluation results before and after the treatment program.

Unique Value: The study will contribute to the literature as it is the first study comparing the superiority of virtual reality training over task-oriented education in individuals with multiple sclerosis and the superiority of virtual reality training and task-oriented education over conventional education. In addition, it will contribute to the literature as it is the first study to observe the effects of task-oriented training and virtual reality training on balance, walking and fatigue in individuals with multiple sclerosis.

DETAILED DESCRIPTION:
Research question or Hypothesis(ies) and Purpose(s):

The aim of the study, which started with the question"Is the effect of virtual reality training on balance, gait and fatigue in individuals with multiple sclerosis superior to task-oriented training?", is to compare the effectiveness of virtual reality training on balance, gait and fatigue in individuals with multiple sclerosis with the effects of task-oriented training.

H0a: Task-oriented training has no effect on balance in individuals with Multiple Sclerosis.

H1a: Task-oriented training has an effect on balance in individuals with Multiple Sclerosis.

H0b: Virtual reality training has no effect on balance in individuals with Multiple Sclerosis.

H1b: Virtual reality training has an effect on balance in individuals with Multiple Sclerosis.

H0c: Task-oriented training has no effect on walking in individuals with Multiple Sclerosis.

H1c: Task-oriented training has an effect on walking in individuals with Multiple Sclerosis H0d: Virtual reality training has no effect on walking in individuals with Multiple Sclerosis H1d: Virtual reality training has an effect on walking in individuals with Multiple Sclerosis.

H0e: Task-oriented training has no effect on fatigue in individuals with Multiple Sclerosis H1e: Task-oriented training has an effect on fatigue in individuals with Multiple Sclerosis.

H0f: Virtual reality training has no effect on fatigue in individuals with Multiple Sclerosis H1f: Virtual reality training has an effect on fatigue in individuals with Multiple Sclerosis.

H0g: Task-oriented training or virtual reality training has no superiority over conventional treatment in individuals with Multiple Sclerosis H1g: Task-oriented training or virtual reality training is superior to conventional treatment in individuals with Multiple Sclerosis.

Type of study:

Randomized controlled trial

Place and time of the research:

It is planned to collect data at Elazig Private Island Special Education and Rehabilitation Center between 15.11.2022 and 15.11.2023.

Population and sample of the research:

The population of the research consists of individuals with MS (Multiple Sclerosis) between the ages of 20-65 at Elazig Private Ada Special Education and Rehabilitation Center. The entire population will be reached among the individuals who agree to participate in the study and who are at Private Ada special education and rehabilitation center located in the center of Elazig, provided that they meet the inclusion criteria. Assignment to groups will be made with a computerized randomizer program. After explaining the purpose and content of the study to individuals, signing the informed consent form, the contact information of those who want to participate voluntarily will be recorded. Individuals will be divided into three groups using the sealed envelope randomization method. They will be randomly assigned to the experimental group, which is the group that will receive task-oriented training, the experimental group, which will be applied Virtual reality training, and the control group, which is the group that will receive conventional treatment.

Inclusion Criteria:

1. Individuals with benign type, relapsing remitting type multiple sclerosis.
2. Individuals between the ages of 20-65.
3. Being between levels 0-5 according to expanded disability status scale (EDSS).
4. Participating in the study voluntarily.

Exclusion Criteria:

1. Having an acute MS attack,
2. Having an orthopedic or systemic problem that will prevent participation in exercises,
3. Having another known neuromuscular disorder other than MS,
4. Having high-level spasticity in the lower extremity (Modified Ashworth Scale score of 3 or 4),
5. Individuals with cardiopulmonary problems that would prevent them from participating in exercise.

Exclusion Criteria:

1. Inability to adapt to treatment sessions.
2. Not attending 25% of treatment sessions
3. Those who experience any health problems during the working period.
4. Those who want to leave the study.
5. Those with vestibular involvement in the virtual reality group.

Study material:

Expanded disability status scale to evaluate physical disability; balance assessment berg balance scale; gait assessment rivermead visual gait assessment scale; Fatigue assessment will be evaluated using the fatigue severity scale. Additionally, Xbox 360 and Kinect® sensor will be used for virtual reality application.

Data collection tools:

Individuals will be evaluated for suitability by a physiotherapist before the preliminary evaluation from the universe of individuals with multiple sclerosis, between the ages of 20-65, at the Private Island Special Education and Rehabilitation Center. Once eligibility is determined, individuals will be assigned to 3 groups. Evaluations will be made one day before the start of the treatment programs for each group and one day after the end of the eight-week treatment program. Individuals' compliance with treatment programs will also be recorded.

Assessment form: Individuals' sociodemographic data will be questioned with the evaluation form. Evaluation form; will question the patient's name-surname, age, gender, height, body weight, and body mass index.

Assessment of Physical Disability: It will be evaluated using the expanded disability status scale. The disability status scale is scored between "0 points" and "10" points. "0-1.5 points" represents normal walking, "8-9.5 points" generally represents wheelchair or bed dependence, and "10 points" represents death due to MS. In other words, as the score increases, the disability rate increases.

Balance Assessment: It will be done using the Berg balance scale. It takes between 15 and 20 minutes to make. The patient who will be evaluated with the Berg balance scale must understand the commands given. 14 basic functions are questioned throughout the evaluation. For example; standing up from a sitting position. Each function is scored with a score between "0" and "4". While a score of 4 indicates that the patient is independent in that function, a score of 0 means that the patient is dependent on that function. 14 basic functions are evaluated throughout the test and the scores given to the patient are collected at the end of the test. As a result, the person evaluated receives a score between 0-56. Scores between 0-20 indicate balance disorder, scores between 21-40 indicate that the balance is acceptable, and scores between 41-56 indicate that the balance is good.

Walking Assessment: Will be evaluated with the Rivermead visual walking assessment scale. In the Rivermead visual gait assessment scale, the upper extremity, stance phase and swing phase are evaluated as separate groups and also questions the individual's use of assistive devices. The scale consists of a total of 20 questions evaluating walking. Each question is generally scored with a score between "0" and "3". "0 points" means normal and "3 points" means severe. As a result, the person evaluated receives a score between 0-59. A high score indicates severe gait disorder.

Fatigue Assessment: Fatigue will be evaluated with the severity scale. The scale consists of 9 questions. Each question consists of 7 points. Each question in the scale is scored between 1 (I completely disagree) and 7 (I completely agree). The lowest score that can be obtained from the scale is 9 and the highest score is 63. The Fatigue Severity Scale is the average of nine sections. A higher score indicates increased fatigue severity. Patients with a Fatigue Severity Scale score less than 4 are considered "not fatigued" and patients with a score greater than 4 are considered "tired".

Variables of the research:

The dependent variables of the research are age, gender, height, weight and body mass index, while the independent variables are balance, walking and fatigue parameters.

Research plan:

The population of the study, planned as a prospective, single-blind randomized controlled study, consists of individuals with MS between the ages of 20-65 at Elazig Private Ada Special Education and Rehabilitation center. For the sample of the study, which is planned to be carried out between 23.09.2022 - 23.09.2024, after the individuals were selected to reach the entire relevant universe, the individuals whose consent form was obtained and who met the inclusion criteria were assigned to the experimental group, the group to be applied task-oriented training with the computerized randomizer program, and the group to be applied virtual reality training to the experimental group. and will be randomly assigned to the control group, which is the group that will receive conventional treatment.

The individuals included in the research will be divided into 3 groups:

1. st Group (experiment): It is planned to provide task-oriented training to the individuals in this group.
2. nd Group (experiment): It is planned to apply virtual reality training to the individuals in this group.
3. rd Group (control): Conventional treatment is planned to be applied to individuals in this group.

The task-oriented training group, which is the experimental group, will be given task-oriented training in the clinic for 40 minutes a day, 3 days a week for 8 weeks. The virtual reality training group will receive virtual reality training for 40 minutes a day, 3 days a week for 8 weeks. The control group will receive conventional treatment 3 days a week for 8 weeks.

Task Oriented Training Procedure;

Task-oriented training focusing on improving balance and walking will consist of 8 different exercise stations. Individuals will continue the exercise at each station for 4 minutes and rest for 1 minute before moving on to the next station. The training completed in this way will consist of a total of 40 minutes and the exercise stations will be applied following the determined order: The exercises will first be demonstrated by the physiotherapist. The aim is to perform exercises at moderate to vigorous intensity. It will be checked that the intensity level of the exercises is moderate and that the perceived effort is 12-15 points according to the Borg Scale. Perception of perceived exertion; It will be controlled by asking to increase the speed, changing the ground, giving double tasks and using obstacles made of wooden blocks. Individuals will be given visual and auditory positive feedback during the exercises.

Sit-stand exercise; sit and stand on chairs of different heights, sit and stand on a exercise ball, sit and stand on a exercise ball with an object in hand.

Get up and walk exercise; walking on different surfaces, walking past obstacles on different surfaces, walking with an object in hand on different surfaces, walking by picking up objects from the ground, walking in a figure of 8 between two chairs.

Walking exercise on sloping ground; Walking on normal inclined ground, walking on soft inclined ground, passing obstacles, walking on soft inclined ground, with an object in hand, passing obstacles.

Step exercise; Step exercise on normal ground, on soft ground, on soft ground with an object in hand.

Stair exercise; climbing up and down steps at different heights. Slalom exercise; Walking between cones at different distances on different surfaces.

Lying exercises; lying forward with feet apart or together in a standing position, reaching forward in a tandem stance.

Balance exercises; Static dynamic balance exercises in single leg and tandem stance.

Virtual Reality Training Procedure;

In general, virtual reality training will be developed taking into account neurorehabilitation principles; Type of game and specificity (there will be exercises specific to the disease), Intensity (will be gradually increased), Progress (exercises will be gradually progressed, variability (the environment will be changed) and Feedback (visual and auditory feedback will be provided). The virtual reality training to be applied will also be fun, It will include attention and problem-solving ability. The difficulty and skill level will gradually increase in order to ensure continuity of motivation and motor learning in individuals. The aim is to perform the exercises at moderate to severe intensity. The intensity level of the exercises should be moderate, and the perceived effort should be 12-15 points according to the Borg Scale. It will be checked upon request.

Participants will be informed about the details of the research to be conducted, and after verbal information about the research protocol to be applied, visual practical training will be given for each test. In the meantime, an adaptation process will be provided by allowing participants to perform the tests in slow forms once. Evaluations will be made one day before the start of the treatment programs for each group and one day after the end of the eight-week treatment program. Individuals' compliance with treatment programs will also be recorded.

Limitations of the research:

One of the limitations of the study is that the universe the investigators created from individuals with multiple sclerosis includes only individuals with benign type and relapsing remitting type multiple sclerosis, and that the results of the study cannot be generalized to other types of MS.

Evaluation of data:

In the power analysis performed before the start of the study, the difference between the Berg balance scale scores in individuals with multiple sclerosis with α = 0.05 and 1-β (power) = 0.80, and the difference between the treatment group (81.9±10.09) and the control group (89.47±6.69) after the study was 7.57 units. Assuming that at least 21 subjects should be included in each group, a total of 63 subjects were calculated. A power analysis was performed to calculate the sample size using the publicly available statistical software Open Source Epidemiologic Statistics for Public Health Version (OpenEpi), version 3 (http://www.openepi.com).

In the study, statistical analysis of the data obtained before and after treatment will be performed with the "Statistical Package for the Social Sciences (SPSS) for Windows Ver 24.0" statistical program. In comparing the pre- and post-treatment data of the treatment groups, Paired T test was used in cases where parametric conditions were met, and Wilcoxon test in non-parametric conditions; In comparing the difference between groups, ANOVA and post-hoc analyzes will be used in cases where parametric conditions are met, and the Kruskal Wallis test will be used in non-parametric cases. In the study, statistical significance (p) will be accepted as being less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with benign type, relapsing remitting type multiple sclerosis.
* Individuals between the ages of 20-65.
* Being between levels 0-5 according to EDSS.
* Participating in the study voluntarily.

Exclusion Criteria:

* Having an acute MS attack,
* Participants have an orthopedic or systemic problem that would prevent them from continuing to exercise,
* Another known neuromuscular disease other than MS,
* Having high-level spasticity (Modified Ashworth Scale score of 3 or 4) in the lower extremity,
* Individuals with cardiopulmonary problems that prevent them from exercising.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Berg Balance Test | 12 weeks
  It takes between 15 and 20 minutes to make. The patient who will be evaluated with the Berg balance scale must understand the commands given. 14 basic functions are questioned throughout the evaluation. For example; standing up from a sitting position. Each function is scored with a score between "0" and "4". While a score of 4 indicates that the patient is independent in that function, a score of 0 means that the patient is dependent on that function. 14 basic functions are evaluated throughout the test and the scores given to the patient are collected at the end of the test. As a result, the person evaluated receives a score between 0-56. Scores between 0-20 indicate balance disorder, scores between 21-40 indicate that the balance is acceptable, and scores between 41-56 indicate that the balance is good.

SECONDARY OUTCOMES:
Fatigue Severity Scale | 12 weeks
  The scale consists of 9 questions. Each question consists of 7 points. Each question in the scale is scored between 1 (I completely disagree) and 7 (I completely agree). The lowest score that can be obtained from the scale is 9 and the highest score is 63. The Fatigue Severity Scale is the average of nine sections. A higher score indicates increased fatigue severity. Patients with a Fatigue Severity Scale score less than 4 are considered "not fatigued" and patients with a score greater than 4 are considered "tired".

OTHER OUTCOMES:
Rivermead Visual Walking Scale | 12 weeks
  In the Rivermead visual gait assessment scale, the upper extremity, stance phase and swing phase are evaluated as separate groups and also questions the individual's use of assistive devices. The scale consists of a total of 20 questions evaluating walking. Each question is generally scored with a score between "0" and "3". "0 points" means normal and "3 points" means severe. As a result, the person evaluated receives a score between 0-59. A high score indicates severe gait disorder.
Expanded Disability Status Scale | 12 weeks
  The disability status scale is scored between "0 points" and "10" points. "0-1.5 points" represents normal walking, "8-9.5 points" generally represents wheelchair or bed dependence, and "10 points" represents death due to MS. In other words, as the score increases, the disability rate increases.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu TALU, Associate Professor, Principal Investigator — Advisor
Locations (1):
- Inonu Univercity, Malatya, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No